CLINICAL TRIAL: NCT00612807
Title: Adapting Marital Therapy in Older Adults With Depression
Brief Title: Treatment of Mood and Marriage Study (TOMMS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00008099; R34MH073677-01A2 (NIH)
Record Dates: First submitted 2008-01-02; First posted 2008-02-12 (Estimated); Results first posted 2011-04-26 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2011-03

CONDITIONS: Major Depressive Disorder; Partner Relational Disorder (V61.10)
Keywords: Older Adults
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Bupropion; Venlafaxine Hydrochloride; Nortriptyline; Tranylcypromine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Medication management with a study doctor every other week.
  Interventions: Drug: As indicated: Sertraline, bupropion, venlafaxine, mirtazepine, nortriptyline, tranylcypromine, lithium augmentation, etc.
- Combination (Experimental): Medication management with a study doctor every other week plus weekly marital therapy.
  Interventions: Behavioral: Weekly marital therapy; Drug: As indicated: Sertraline, bupropion, venlafaxine, mirtazepine, nortriptyline, tranylcypromine, lithium augmentation, etc.

INTERVENTIONS:
Behavioral: Weekly marital therapy — Weekly marital therapy for 6 months.
  Other Names: Integrative Behavioral Couple Therapy
  Arms: Combination
Drug: As indicated: Sertraline, bupropion, venlafaxine, mirtazepine, nortriptyline, tranylcypromine, lithium augmentation, etc. — Study doctor may prescribe antidepressant medication for the treatment of depression. Medications will be prescribed according to empirically supported guidelines outlined in the Duke Somatic Treatment Algorithm for Geriatric Depression (STAGED Approach; Steffens, 2002).
  SSRIs (daily dose of at least 20 mg for citalopram, 20 mg for fluoxetine, 100 mg for sertraline, 20 mg for paroxetine)
  SNRIs (e.g., venlafaxine)
  Bupropion SR (achieve dose of at least 150 mg BID)
  Mirtazapine
  Tricyclic antidepressants (nortriptyline with drug levels 80-120 ng/dl)
  Lithium augmentation
  MAOI (daily dose of at least 30 mg tranylcypromine or 45 mg of phenelzine)

SUMMARY:
The primary goal of this study is to develop and test a depression-specific marital therapy tailored for use with older adult populations.

DETAILED DESCRIPTION:
Major depression has been associated with many individual and interpersonal problems in later life, including inadequate social support, marital distress, spousal depression, poor physical health, and higher rates of mortality. Marital therapy has shown promise as a treatment for depression and coexisting marital distress in younger cohorts, and there is a robust association between social support and depressive symptoms in older adults. The combination of couple therapy and antidepressant medication may provide an ideal treatment for older adults by targeting interpersonal and biochemical aspects of depression.

Couples interested in this study will complete an initial assessment with study personnel. In Phase I, eligible couples will receive weekly marital therapy and the depressed partner will receive medication management with a study doctor for 6 months. In Phase II, couples will be randomly assigned to either the combination treatment (marital therapy plus medication management) or medication management alone for 6 months. At the end of the treatment phase, a thorough assessment will be completed. A follow-up assessment will be completed 6 months after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* One partner must receive a clinical diagnosis of major depressive disorder based upon our assessment
* Couples must be living together
* Either partner must report marital distress or tension
* Willing to take antidepressant medication and participate in weekly marital therapy and assessments
* The depressed partner cannot be involved in any other psychosocial treatment
* Score above 24 on the Mini Mental Status Exam

Exclusion Criteria:

* Both partners meet diagnostic criteria for major depressive disorder based on our evaluation
* Coexisting bipolar or psychotic disorder
* Evidence of a primary substance abuse or dependence disorder
* Current ECT treatment
* Evidence of active and severe domestic violence

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill S. Compton, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Child & Family Studies Center; Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Futterman A, Gallagher D, Thompson LW, Lovett S, Gilewski M. Retrospective assessment of marital adjustment and depression during the first 2 years of spousal bereavement. Psychol Aging. 1990 Jun;5(2):277-83. doi: 10.1037//0882-7974.5.2.277. PMID 2378693
- [Background] Jacobson, N.S. & Christensen, A. (1996). Acceptance and Change in Couple Therapy: A Therapist's Guide to Transforming Relationships. New York: W.W. Norton & Company, Inc.
- [Background] Oxman TE, Berkman LF, Kasl S, Freeman DH Jr, Barrett J. Social support and depressive symptoms in the elderly. Am J Epidemiol. 1992 Feb 15;135(4):356-68. doi: 10.1093/oxfordjournals.aje.a116297. PMID 1550090
- [Background] Tower RB, Kasl SV. Depressive symptoms across older spouses and the moderating effect of marital closeness. Psychol Aging. 1995 Dec;10(4):625-38. doi: 10.1037//0882-7974.10.4.625. PMID 8749590
- [Background] Gerson S, Belin TR, Kaufman A, Mintz J, Jarvik L. Pharmacological and psychological treatments for depressed older patients: a meta-analysis and overview of recent findings. Harv Rev Psychiatry. 1999 May-Jun;7(1):1-28. PMID 10439302
- [Background] Murrell SA, Himmelfarb S, Wright K. Prevalence of depression and its correlates in older adults. Am J Epidemiol. 1983 Feb;117(2):173-85. doi: 10.1093/oxfordjournals.aje.a113528. PMID 6829547
- [Background] Simons AD, Murphy GE, Levine JL, Wetzel RD. Cognitive therapy and pharmacotherapy for depression. Sustained improvement over one year. Arch Gen Psychiatry. 1986 Jan;43(1):43-8. doi: 10.1001/archpsyc.1986.01800010045006. PMID 3942473
- [Background] Baldessarini RJ. Current status of antidepressants: clinical pharmacology and therapy. J Clin Psychiatry. 1989 Apr;50(4):117-26. PMID 2647712
- [Background] Scogin F, McElreath L. Efficacy of psychosocial treatments for geriatric depression: a quantitative review. J Consult Clin Psychol. 1994 Feb;62(1):69-74. doi: 10.1037//0022-006x.62.1.69. PMID 8034832
- [Background] Thase ME, Greenhouse JB, Frank E, Reynolds CF 3rd, Pilkonis PA, Hurley K, Grochocinski V, Kupfer DJ. Treatment of major depression with psychotherapy or psychotherapy-pharmacotherapy combinations. Arch Gen Psychiatry. 1997 Nov;54(11):1009-15. doi: 10.1001/archpsyc.1997.01830230043006. PMID 9366657
- [Background] Reynolds CF 3rd, Frank E, Perel JM, Imber SD, Cornes C, Miller MD, Mazumdar S, Houck PR, Dew MA, Stack JA, Pollock BG, Kupfer DJ. Nortriptyline and interpersonal psychotherapy as maintenance therapies for recurrent major depression: a randomized controlled trial in patients older than 59 years. JAMA. 1999 Jan 6;281(1):39-45. doi: 10.1001/jama.281.1.39. PMID 9892449
- [Background] Holahan CJ, Moos RH. Social support and psychological distress: a longitudinal analysis. J Abnorm Psychol. 1981 Aug;90(4):365-70. doi: 10.1037//0021-843x.90.4.365. No abstract available. PMID 7264067
- [Background] George LK, Blazer DG, Hughes DC, Fowler N. Social support and the outcome of major depression. Br J Psychiatry. 1989 Apr;154:478-85. doi: 10.1192/bjp.154.4.478. PMID 2590779
- [Background] Levenson RW, Carstensen LL, Gottman JM. The influence of age and gender on affect, physiology, and their interrelations: a study of long-term marriages. J Pers Soc Psychol. 1994 Jul;67(1):56-68. doi: 10.1037//0022-3514.67.1.56. PMID 8046584
- [Background] Jacobson NS, Holtzworth-Munroe A, Schmaling KB. Marital therapy and spouse involvement in the treatment of depression, agoraphobia, and alcoholism. J Consult Clin Psychol. 1989 Feb;57(1):5-10. doi: 10.1037//0022-006x.57.1.5. PMID 2647802
- [Background] O'Leary, KD, Christian, JL, & Mendell, NR (1994). A closer look at the link between marital discord and depressive symptomatology. Journal of Social and Clinical Psychology, 13, 33-41.
- [Background] Jacobson NS, Dobson K, Fruzzetti AE, Schmaling KB, Salusky S. Marital therapy as a treatment for depression. J Consult Clin Psychol. 1991 Aug;59(4):547-57. doi: 10.1037//0022-006x.59.4.547. PMID 1918559
- [Background] Jacobson NS, Fruzzetti AE, Dobson K, Whisman M, Hops H. Couple therapy as a treatment for depression: II. The effects of relationship quality and therapy on depressive relapse. J Consult Clin Psychol. 1993 Jun;61(3):516-9. doi: 10.1037//0022-006x.61.3.516. PMID 8326054
- [Background] O'Leary KD, Beach SR. Marital therapy: a viable treatment for depression and marital discord. Am J Psychiatry. 1990 Feb;147(2):183-6. doi: 10.1176/ajp.147.2.183. PMID 2301656
- [Background] Leff J, Vearnals S, Brewin CR, Wolff G, Alexander B, Asen E, Dayson D, Jones E, Chisholm D, Everitt B. The London Depression Intervention Trial. Randomised controlled trial of antidepressants v. couple therapy in the treatment and maintenance of people with depression living with a partner: clinical outcome and costs. Br J Psychiatry. 2000 Aug;177:95-100. doi: 10.1192/bjp.177.2.95. PMID 11026946
- [Background] Jacobson NS, Christensen A, Prince SE, Cordova J, Eldridge K. Integrative behavioral couple therapy: an acceptance-based, promising new treatment for couple discord. J Consult Clin Psychol. 2000 Apr;68(2):351-5. doi: 10.1037//0022-006x.68.2.351. PMID 10780137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Older, maritally-distressed couples with a depressed spouse were recruited via flyers and referral for participation in a study on couples therapy in older adults. Recruitment for Phase I occurred from 10/2006 to 5/2007; recruitment for Phase II occurred from 7/2007 to 5/2009.
Pre-assignment Details: No participants who met eligibility criteria were excluded before assignment to treatment condition.
Groups:
- Semi-weekly Medication Management: Medication management with a study doctor every other week.
- Semi-weekly Medication Management + Weekly Marital Therapy: Medication management with a study doctor every other week plus weekly marital therapy.
Period: Overall Study
Arm/Group | Semi-weekly Medication Management | Semi-weekly Medication Management + Weekly Marital Therapy
Started | 14 | 28
Completed | 12 | 28
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semi-weekly Medication Management | Semi-weekly Medication Management + Weekly Marital Therapy | Total
Number analyzed (Participants) | 14 | 28 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 10 | 13
  >=65 years | 11 | 18 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 71.2 (6.0) | 67.2 (7.5) | 68.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 7 | 14 | 21
Region of Enrollment [Number; unit: participants]
  United States | 14 | 28 | 42

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS)
Description: The HDRS is a semi-structured interview administered by a trained independent evaluator, and used for rating the severity of depressive symptoms. Scores range from 0 to 50, with higher scores indicating greater severity of depression.
Time Frame: pre-treatment, monthly, post-treatment, 6 month follow-up
Measure: Mean (Standard Deviation); unit: Score on HDRS
Arm/Group | Semi-weekly Medication Management | Semi-weekly Medication Management + Weekly Marital Therapy
Number analyzed (Participants) | 14 | 28
Score on HDRS
  Baseline assessment (Depressed spouse) | 17.86 (2.11) | 19.0 (3.80)
  Post-test assessment (Depressed spouse) | 5.00 (5.44) | 7.29 (5.13)
  Follow-up assessment (Depressed spouse) | 9.17 (7.52) | 8.14 (5.76)
  Baseline assessment (Non-depressed spouse) | 5.14 (3.76) | 8.86 (5.04)
  Post-test assessment (Non-depressed spouse) | 5.33 (6.56) | 3.29 (2.67)
  Follow-up assessment (Non-depressed spouse) | 3.83 (2.99) | 5.71 (4.06)
Statistical Analysis 1: Comparison: Semi-weekly Medication Management vs Semi-weekly Medication Management + Weekly Marital Therapy; Utilized a hierarchical linear model with time nested within individual and individual nested within couple. Given the small sample size, we chose to include participants' baseline depression scores as a covariate, and model the trajectory of change in depression scores beginning with the second assessment, which occurred one month into the study. Additional fixed effect predictors included status as identified patient or spouse, treatment condition, time, and all possible interactions; Test type: Non-Inferiority or Equivalence — Testing whether slope of change over time varied by identified patient status and treatment condition; p = 0.056, Fixed effect in multi-level model — Interaction indicates that slope of change varied by identified patient status and tx condition. Slope of change in depression was significantly negative for everyone but identified patients in the control condition; Interaction term = -0.56, Standard Error of Mean 0.29

2. Primary Outcome: Dyadic Adjustment Scale (DAS)
Description: The DAS is a self-report measure of marital adjustment that includes questions about agreement on lifestyle and household decisions, level of conflict, level of cooperation, and affection. Scores range from 0 to 151, with higher scores representing better relationship functioning.
Time Frame: pre-treatment, monthly, post-treatment, 6 month follow-up
Measure: Mean (Standard Deviation); unit: Score on DAS measure
Arm/Group | Semi-weekly Medication Management | Semi-weekly Medication Management + Weekly Marital Therapy
Number analyzed (Participants) | 14 | 28
Score on DAS measure
  Baseline assessment (Depressed spouse) | 72.14 (24.30) | 84.43 (11.89)
  Post-test assessment (Depressed spouse) | 84.17 (23.17) | 92.27 (16.27)
  Follow-up assessment (Depressed spouse) | 89.67 (24.23) | 91.07 (19.85)
  Baseline assessment (Non-depressed spouse) | 91.0 (18.32) | 88.29 (15.46)
  Post-test assessment (Non-depressed spouse) | 93.33 (29.75) | 97.57 (17.49)
  Follow-up assessment (Non-depressed spouse) | 104.17 (13.76) | 98.31 (20.52)
Statistical Analysis 1: Comparison: Semi-weekly Medication Management vs Semi-weekly Medication Management + Weekly Marital Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Testing whether slope of change over time varied by identified patient status and treatment condition; p = 0.32, Fixed effect in multi-level model; Interaction term = 0.64, Standard Error of Mean 0.65
Statistical Analysis 2: Comparison: Semi-weekly Medication Management vs Semi-weekly Medication Management + Weekly Marital Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Testing whether means at each timepoint varied by identified patient status and treatment condition; p = 0.005, Fixed effect in multi-level model — We probed this interaction and discovered that at each assessment, spouses in the couple therapy + medication treatment group reported greater dyadic adjustment than did spouses in the medication alone condition (b = 10.53, z = 2.72, p = 0.006); Interaction term = -12.97, Standard Error of Mean 4.52

3. Secondary Outcome: Frequency & Acceptability of Partner Behavior
Time Frame: Pre-treatment, post-treatment, 6 month follow-up
Reporting Status: Not Posted

4. Secondary Outcome: Conflict Tactics Scale
Time Frame: pre-treatment, post-treatment, 6 month follow-up
Reporting Status: Not Posted

5. Secondary Outcome: SCID Mood Disorders
Time Frame: pre-treatment, post-treatment, 6 month follow-up
Reporting Status: Not Posted

6. Secondary Outcome: Personal Assessment of Intimacy in Relationships
Time Frame: pre-treatment, post-treatment, 6 month-followup
Reporting Status: Not Posted

7. Secondary Outcome: Beck Anxiety Inventory
Time Frame: pre-treatment, post-treatment, 6 month follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Semi-weekly Medication Management | Semi-weekly Medication Management + Weekly Marital Therapy
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/28
Other Adverse Events (participants affected / at risk) | 0/14 | 2/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semi-weekly Medication Management (N=14) | Semi-weekly Medication Management + Weekly Marital Therapy (N=28)
Passive suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) — Passive suicidal ideation without intent to act.

LIMITATIONS AND CAVEATS:
Small sample size limits power to detect differences. Some participants reported difficulty understanding how to complete the questions, which may introduce additional variability into the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No